CLINICAL TRIAL: NCT04014907
Title: Open Repair Versus Branched Endograft Repair for Treatment of Residual Chronic Aortic Arch Dissection During Follow-up After Open Type A Acute Ascending Aorta Replacement: Results From an International Multicenter Study.
Status: Completed | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, TINELLI GIOVANNI, Head of the Endovascular Therapies Unit, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 15530/19
Record Dates: First submitted 2019-07-09; First posted 2019-07-10 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Peri-operative Mortality

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Frozen Elephant Trunk Technique — Endovascular technique forTAA repair

SUMMARY:
This study aims to evaluate peri-operative mortality and main post-operative complications (for example cardiovascular, respiratory and renal) in patients treated with frozen elephant trunk techinque.

ELIGIBILITY:
Inclusion Criteria:

* patients with post-dissection arch aneurysm with a maximal aortic diameter >55mm or rapid growth (>10mm/year)

Exclusion Criteria:

* Emergency setting

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients undergoing endovascular TAA repair with Frozen Elephant Trunk Technique
Sampling Method: Non-Probability Sample
Enrollment: 170 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Peri-operatory mortality | 36 months

SECONDARY OUTCOMES:
Post-operatory complications | 36 months

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Universitario A. Gemelli IRCCS, Roma, RM, Italy